CLINICAL TRIAL: NCT00003881
Title: Phase II Pilot Trial of Carboplatin, Paclitaxel, and Herceptin in HER2/Neu (+) Advanced NSCLC
Brief Title: Trastuzumab Plus Chemotherapy in Treating Patients With Advanced Non-small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eastern Cooperative Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000067048; ECOG-2598
Record Dates: First submitted 1999-11-01; First posted 2004-07-19 (Estimated); Last update posted 2013-06-21 (Estimated); Status verified 2004-03

CONDITIONS: Lung Cancer
Keywords: recurrent non-small cell lung cancer; stage IIIB non-small cell lung cancer; stage IV non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Trastuzumab; Carboplatin; Paclitaxel

INTERVENTIONS:
Biological: trastuzumab
Drug: carboplatin
Drug: paclitaxel

SUMMARY:
RATIONALE: Monoclonal antibodies can locate tumor cells and either kill them or deliver tumor-killing substances to them without harming normal cells. Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining monoclonal antibody therapy with chemotherapy may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of the monoclonal antibody trastuzumab plus carboplatin and paclitaxel in treating patients who have advanced non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Assess the toxicity of monoclonal antibody HER2 with carboplatin and paclitaxel in patients with HER2 positive non-small cell lung cancer. II. Determine median time to progression and one year freedom from progression in this patient population. III. Evaluate one year survival rate and overall objective response rate in this patient population.

OUTLINE: Patients receive paclitaxel IV over 3 hours immediately followed by carboplatin IV over 30 minutes immediately followed by monoclonal antibody HER2 IV over 30-90 minutes on day 1. Patients also receive monoclonal antibody HER2 on days 8 and 15. Treatment is repeated every 3 weeks for 6 courses. After 6 courses of treatment, patients may receive monoclonal antibody HER2 weekly for up to 1 year in the absence of disease progression or unacceptable toxicity. Patients are followed every 3 months for 2 years, every 6 months for 3 years and once a year thereafter until disease progression or death.

PROJECTED ACCRUAL: A total of 22-44 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed non-small cell lung cancer (NSCLC) Recurrent AND/OR Stage IIIB with pleural or pericardial effusion OR Stage IV Must have at least one bidimensionally measurable lesion Must be HER2 positive (1-3+) Brain metastases allowed, if symptoms controlled and not requiring steroids Prior/Concurrent Therapy-- Biologic therapy: Not specified Chemotherapy: No prior chemotherapy for NSCLC Endocrine therapy: No concurrent steroids Radiotherapy: At least 2 weeks since prior radiotherapy Surgery: Not specified

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: ECOG 0-1 Life expectancy: Not specified Hematopoietic: Absolute neutrophil count at least 1,500/mm3 Platelet count at least 100,000/mm3 Hepatic: Bilirubin no greater than 1.5 mg/dL Transaminases no greater than 5 times upper limit of normal Renal: Creatinine no greater than 2 mg/dL Cardiovascular: No uncontrolled angina pectoris and arrhythmias No myocardial infarction within past 3 months No uncompensated congestive heart failure Ejection fraction at least 45% Other: No active infections Not pregnant or nursing Fertile patients must use effective contraception HIV negative No other active malignancies No evidence of peripheral sensory neuropathy of at least grade 2

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1999-05; Study Completion 2004-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Corey J. Langer, MD, Study Chair — Fox Chase Cancer Center
Locations (71):
- United States (68):
  - CCOP - Scottsdale Oncology Program, Scottsdale, Arizona
  - Beckman Research Institute, City of Hope, Los Angeles, California
  - Veterans Affairs Medical Center - Palo Alto, Palo Alto, California
  - Stanford University Medical Center, Stanford, California
  - CCOP - Colorado Cancer Research Program, Inc., Denver, Colorado
  - CCOP - Christiana Care Health Services, Wilmington, Delaware
  - Walter Reed Army Medical Center, Washington D.C., District of Columbia
  - Veterans Affairs Medical Center - Gainsville, Gainesville, Florida
  - Sylvester Cancer Center, University of Miami, Miami, Florida
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Veterans Affairs Medical Center - Tampa (Haley), Tampa, Florida
  - Emory University Hospital - Atlanta, Atlanta, Georgia
  - Veterans Affairs Medical Center - Atlanta (Decatur), Decatur, Georgia
  - Robert H. Lurie Comprehensive Cancer Center, Northwestern University, Chicago, Illinois
  - Veterans Affairs Medical Center - Chicago (Lakeside), Chicago, Illinois
  - CCOP - Central Illinois, Decatur, Illinois
  - CCOP - Evanston, Evanston, Illinois
  - CCOP - Illinois Oncology Research Association, Peoria, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - Indiana University Cancer Center, Indianapolis, Indiana
  - Veterans Affairs Medical Center - Indianapolis (Roudebush), Indianapolis, Indiana
  - CCOP - Cedar Rapids Oncology Project, Cedar Rapids, Iowa
  - CCOP - Iowa Oncology Research Association, Des Moines, Iowa
  - CCOP - Wichita, Wichita, Kansas
  - MBCCOP - LSU Medical Center, New Orleans, Louisiana
  - CCOP - Ochsner, New Orleans, Louisiana
  - Johns Hopkins Oncology Center, Baltimore, Maryland
  - New England Medical Center Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - CCOP - Ann Arbor Regional, Ann Arbor, Michigan
  - CCOP - Kalamazoo, Kalamazoo, Michigan
  - CCOP - Duluth, Duluth, Minnesota
  - Veterans Affairs Medical Center - Minneapolis, Minneapolis, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - CCOP - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - CCOP - Southern Nevada Cancer Research Foundation, Las Vegas, Nevada
  - Veterans Affairs Medical Center - East Orange, East Orange, New Jersey
  - CCOP - Northern New Jersey, Hackensack, New Jersey
  - Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Veterans Affairs Medical Center - Albany, Albany, New York
  - Veterans Affairs Medical Center - Brooklyn, Brooklyn, New York
  - Veterans Affairs Medical Center - New York, New York, New York
  - Kaplan Cancer Center, New York, New York
  - University of Rochester Cancer Center, Rochester, New York
  - Albert Einstein Comprehensive Cancer Center, The Bronx, New York
  - CCOP - Merit Care Hospital, Fargo, North Dakota
  - Ireland Cancer Center, Cleveland, Ohio
  - Veterans Affairs Medical Center - Cleveland, Cleveland, Ohio
  - CCOP - Columbus, Columbus, Ohio
  - CCOP - Toledo Community Hospital Oncology Program, Toledo, Ohio
  - CCOP - St. Francis Hospital/Natalie Warren Bryant Cancer Center, Tulsa, Oklahoma
  - CCOP - Geisinger Clinical and Medical Center, Danville, Pennsylvania
  - Allegheny University Hospitals- Hahnemann, Philadelphia, Pennsylvania
  - University of Pennsylvania Cancer Center, Philadelphia, Pennsylvania
  - Kimmel Cancer Center of Thomas Jefferson University - Philadelphia, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - University of Pittsburgh Cancer Institute, Pittsburgh, Pennsylvania
  - Veterans Affairs Medical Center - Pittsburgh, Pittsburgh, Pennsylvania
  - CCOP - MainLine Health, Wynnewood, Pennsylvania
  - CCOP - Sioux Community Cancer Consortium, Sioux Falls, South Dakota
  - Veterans Affairs Medical Center - Nashville, Nashville, Tennessee
  - Vanderbilt Cancer Center, Nashville, Tennessee
  - Veterans Affairs Medical Center - Madison, Madison, Wisconsin
  - University of Wisconsin Comprehensive Cancer Center, Madison, Wisconsin
  - CCOP - Marshfield Medical Research and Education Foundation, Marshfield, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - Veterans Affairs Medical Center - Milwaukee (Zablocki), Milwaukee, Wisconsin
- Puerto Rico (2):
  - MBCCOP - San Juan, San Juan
  - Veterans Affairs Medical Center - San Juan, San Juan
- Pretoria Academic Hospital, Pretoria, South Africa

REFERENCES:
- [Result] Langer CJ, Stephenson P, Thor A, Vangel M, Johnson DH; Eastern Cooperative Oncology Group Study 2598. Trastuzumab in the treatment of advanced non-small-cell lung cancer: is there a role? Focus on Eastern Cooperative Oncology Group study 2598. J Clin Oncol. 2004 Apr 1;22(7):1180-7. doi: 10.1200/JCO.2004.04.105. Epub 2004 Feb 23. PMID 14981103
- [Result] Huang C, Stephenson P, Langer CJ, et al.: Trastuzumab in combination with paclitaxel/carboplatin in advanced non-small cell lung cancer: final report of ECOG 2598. [Abstract] Lung Cancer 41 (Suppl 2): A-P628, S251, 2003.
- [Result] Schiller J, Langer CJ, Thor A, et al.: Trastuzumab in combination with paclitaxel/carboplatin advanced non-small cell lung cancer: final report of ECOG 2598. [Abstract] Proceedings of the American Society of Clinical Oncology 22: A-2606, 2003.
- [Result] Langer CJ, Adak S, Thor A, et al.: Phase II Eastern Cooperative Oncology Group (ECOG) pilot study of paclitaxel (P), carboplatin (C), and trastuzumab (T) in HER-2/neu (+) advanced non-small cell lung cancer (NSCLC): early analysis of E2598. [Abstract] Proceedings of the American Society of Clinical Oncology 20: A-1257, 2001.